CLINICAL TRIAL: NCT03013231
Title: Effect of Patient Resilience on Return to Sport Post ACL Reconstruction Surgery
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Scott Kaar, MD, Associate Professor, Dept. of Orthopaedic Surgery, St. Louis University
Other Study IDs: 47659; 27659 (Other: SLU IRB)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: ACL Reconstruction; Return to Sport; Resilience
MeSH Terms: interventions — The Brief Resilience Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- s/p ACLR: Patients having undergone ACL Reconstruction Surgery with goal of returning to sport. 6 months post-op, patients will complete the BRS survey as a method of evaluating resilience.
  Interventions: Behavioral: Brief Resilience Scale

INTERVENTIONS:
Behavioral: Brief Resilience Scale — 6 months post-op, patients will complete the BRS survey as a method of evaluating resilience.
  Other Names: BRS

SUMMARY:
Despite the large majority of patients that undergo ACL reconstruction reporting successful outcomes in regard to tests of knee function, only about 2/3 return to their prior level or athletic activity after surgery. A large amount of research has been conducted investigating the effects of psychological factors on return to sports after ACL reconstruction; however, the specific role of resilience has yet to be solely analyzed. This study aims to determine the effect of variations in patient resilience on their return to sports after surgery.

DETAILED DESCRIPTION:
Meta-analysis of post ACL reconstruction return to sport suggests that despite approximately 90% of patients achieving successful outcomes in terms of objectively measurable knee function, only 63% return to their pre-injury sport participation rate. This leads one to question what factors other than knee function may contribute to such a discrepancy. Prior studies have shown psychological factors, such as fear of re-injury, can play in role in whether a patient returns to play. However, the role of patient resilience on recovery is less clear. This research will examine the effect of patient resilience on post-ACLR return to sport. The Brief Resiliency Scale (BRS), a proven method of assessing ability to recover from stressful situations, will be used to evaluate patient resilience. The role of resilience on recovery post shoulder surgery, as well as rehabilitation in post-operative orthopaedic geriatric patients has been examined; however, the effect of resilience on specifically ACLR return to sport has yet to be studied.

This research will provide insight as to how to identify patients at high risk for not returning to sport, the first step in improving return to sport outcomes in ACL reconstruction patients.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients
* Isolated ACL tear having undergone surgical reconstruction.

Exclusion Criteria:

* Non-English speaking patients.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: English speaking patients 14 yrs of age or older with isolated ACL tear and having undergone surgical reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Return to Sport | 1 year
  Whether the patient has returned to sport s/p ACLR

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kaar, MD, Principal Investigator — St. Louis University
Locations (1):
- SSM Health Saint Louis University Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313